CLINICAL TRIAL: NCT07340827
Title: A Parallel-group Treatment, 2-arm Study to Compare the Efficacy and Safety of Follitropin Alfa and Lutropin Alfa Fixed Dose Combination Versus hMG for Inducing Follicular Development in Japanese Participants With LH and FSH Deficiency Undergoing ART
Brief Title: A Study to Compare the Efficacy and Safety of Follitropin Alfa/Lutropin Alfa Versus hMG in Japanese Participants With LH and FSH Deficiency Undergoing ART (HINATA)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS132705_0007
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Infertility
Keywords: Gonadotropins, infertility, prefilled pen
MeSH Terms: conditions — Infertility | interventions — cetrorelix; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Follitropin alfa/lutropin alfa (Experimental): Participants will receive fixed combination product of recombinant Follitropin alfa (rechFSH)/lutropin alfa (rechLH) in a 2:1 ratio.
  Interventions: Combination Product: Follitropin alfa/lutropin alfa (MBJ-0011); Drug: Cetrorelix acetate; Drug: Coriogonadotropin alfa; Drug: Progesterone gel
- Arm 2: Human Menopausal Gonadotropin (hMG) (Active Comparator)
  Interventions: Drug: hMG; Drug: Cetrorelix acetate; Drug: Coriogonadotropin alfa; Drug: Progesterone gel

INTERVENTIONS:
Combination Product: Follitropin alfa/lutropin alfa (MBJ-0011) — Follitropin alfa and lutropin alfa will be administered subcutaneously once daily with a starting dose of 150 International Unit (IU) of follitropin alfa, 75 IU of lutropin alfa, in ovarian stimulation up to 18 days.
  Other Names: MBJ-0011; r-hFSH/r-hLH
  Arms: Arm 1: Follitropin alfa/lutropin alfa
Drug: hMG — Participants will receive 150 IU as solvent, subcutaneously, for solution for injection, daily (up to 18 days) during ovarian stimulation.
  Arms: Arm 2: Human Menopausal Gonadotropin (hMG)
Drug: Cetrorelix acetate — Participants will receive 250 micrograms (mcg) of Cetrorelix acetate as Powder for reconstitution to a solution for injection with diluent in ampule, daily from Day 5 or 6 of stimulation up to the day of r-hCG.
  Other Names: GnRH; antagonist
Drug: Coriogonadotropin alfa — Participants will receive 250 mcg of r-hCG, as solution for injection, subcutaneously, during final follicular maturation.
  Other Names: r-hCG
Drug: Progesterone gel — Participants will self-administer progesterone gel 8 percent, with an applicator, at a dose of 90 milligram (mg), intravaginally, daily from oocyte retrieval during Luteal phase support.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of follitropin alfa/lutropin alfa in Japanese participants with Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) deficiency undergoing Assisted reproductive technology (ART).

The study duration is approximately 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy in Part A.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are premenopausal wishing to conceive
* Participants with maximum 1 previous stimulation for assisted reproductive technology (ART) without pregnancy
* Japanese Participants
* Participants are women with Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) deficiency congenital or acquired
* Participants have a vaginal ultrasound scan showing both ovaries and no clinically significant uterine abnormality and a normal antral follicle count (AFC) of at least 5 follicles 2 to 10 millimeter (mm) in diameter per ovary
* A semen analysis of the male partner been performed within 3 months prior to signature of informed consent and suitable for assisted reproductive technology
* Participants have a normal cervical ThinPrep® cytologic test, (TCT) or Pap smear within 12 months of Screening. If not available, a cervical smear will be performed as part of screening
* Other protocol defined criteria may apply

Exclusion Criteria:

* Participants with history of severe OHSS in any previous ovarian stimulation cycle
* Participants with Polycystic ovarian syndrome (PCOS) according to Rotterdam modified definition
* Participants with contraindication to treatment with gonadotropins, hypersensitivity to gonadotropins or to any of the excipients
* Participants with presence of known or suspected gonadotropin- or estrogen dependent malignancy (example. ovarian-, uterine-, or mammary carcinoma)
* Participants with ovarian enlargement or cyst of unknown etiology, or presence of an ovarian cyst greater than 25 millimeters before Day 1
* other protocol defined exclusion criteria may apply

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Total number of oocytes retrieved | At approximately 36 to 38 hours after r-hCG administration (Day 4)
  Mean number of oocytes retrieved will be calculated. Oocyte retrieval was a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.

SECONDARY OUTCOMES:
Total dose of gonadotropin (IU) used | At Visit 3 after ovarian stimulation from Day 5 until Day of r-hCG (maximum 18 days)
  Total dose of Human Menopausal Gonadotropin (hMG) referred as IU of FSH.
Number of Days of Gonadotropin Treatment | At Visit 3 after ovarian stimulation from Day 5-18
  Total number of days of ovarian stimulation will be reported.
Total Number of Follicles Measuring greater than or equal to 14 millimeter (mm) and greater than or equal to 17 mm in diameter | During Ovarian stimulation (Day 5 to Day 18)
Serum Estradiol (E2) levels | At Visit 3 after ovarian stimulation from Day 5-18
Proportion of 2 Pronuclei Embryos/Fertilized Oocytes | At 18 (Plus or minus two hours) hours after insemination
  The proportion of oocytes that fertilized after they were inseminated with the sperm will be reported.
Number of blastocysts frozen | 5 days after insemination
  After the transfer of 1 fresh blastocysts - spare ones will be frozen.
Number of Participants With Clinical Pregnancy | 35-42 days after Visit 5 (Blastocyst transfer)
  A clinical pregnancy is a pregnancy that is confirmed by both pregnancy test (beta-hCG test) and sonographic confirmation of a gestational sac or with or without heartbeat (fetal sac).
Number of Participants With Ongoing Pregnancy | up to 80 days after blastocyst transfer (pregnancy week 11 to 12)
  Ongoing pregnancy will be confirmed with transvaginal ultrasound (TVUS) showing heartbeat.
Number of Participants With Treatment-Emergent Adverse Events and Treatment related Adverse Events | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
Number of Participants With Ovarian Hyperstimulation Syndrome (OHSS) | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
Number of Participants With Mild, Moderate, and Severe Ovarian Hyperstimulation Syndrome | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
Number of Cycles Cancelled due to Risk of Ovarian Hyperstimulation Syndrome | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
Number of Participants With Clinically Significant Changes in Laboratory Parameters and Vital Signs | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
Number of Participants Experiencing Local Reactions | 5.5 months for nonpregnant participants and 13 months for participants with confirmed pregnancy
  Pain redness, swelling, bruising, and itching around the injection site will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union.
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/_en
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html